CLINICAL TRIAL: NCT00983827
Title: Safety and Efficacy of Aquatic Treadmill Therapy for Improving Economy of Gait, Gait Speed, Balance, Cardiovascular Fitness, and Quality of Life in Ambulatory Adult Stroke Patients: A Pilot Study
Brief Title: Aquatic Treadmill Therapy for Improving Gait, Balance, Fitness and Quality of Life in Stroke Patients
Acronym: ATT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Steven Edgley, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 28376; ATT-01
Record Dates: First submitted 2009-08-25; First posted 2009-09-24 (Estimated); Results first posted 2013-01-15 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2012-12

CONDITIONS: Ischemic or Hemorrhagic Stroke; Hemiparesis
MeSH Terms: conditions — Ischemia; Hemorrhagic Stroke; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aquatic treadmill training (Experimental): Aquatic treadmill training (ATT) is a pool-based treadmill training that combines the three concepts of unweighting the body, treadmill training, and the resistance effects of water into one modality.
  Interventions: Device: Aquatic treadmill training

INTERVENTIONS:
Device: Aquatic treadmill training — HydroWorx aquatic therapy pool with an underwater, integrated and adjustable speed treadmill

SUMMARY:
This study aims to determine if Aquatic Treadmill Therapy is effective for improving economy of gait, gait speed, balance, and cardiovascular fitness in people with chronic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with ischemic or hemorrhagic stroke with hemiparesis who have chronic deficits in gait, falls and/or poor fitness

Exclusion Criteria:

* Subjects with medical co-morbidities that may affect gait and endurance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, PM&R Division, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aquatic Treadmill Training
Started | 8
Completed | 7
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Aquatic Treadmill Training
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 53.5 (6.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Safety
Description: Number of procedure related adverse events that occurred during study.
Time Frame: 16 weeks
Measure: Number; unit: adverse events
Arm/Group | Aquatic Treadmill Training
Number analyzed (Participants) | 8
adverse events | 0

ADVERSE EVENTS:
Arm/Group | Aquatic Treadmill Training
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aquatic Treadmill Training (N=8)
Sharp Head Pain (General disorders) | 1 (1) — Event determined not to be related to research.
Fall (Injury, poisoning and procedural complications) | 1 (1) — Event determined not to be related to research.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes